Official Title: The Impact of Cannabidiol (CBD) Health Claims at Point-of-Sale on Consumer

Perceptions and Behavior: Online Survey

NCT06069713

IRB-Approved Date: 7/27/2023

## Consent

The Impact of Cannabidiol (CBD) Health Claims at Point-of-Sale on Consumer Perceptions and Behavior Aim 2: Consumer Perception Survey

## Wake Forest Health Survey

You are eligible to complete a survey as part of a research study being conducted by Wake Forest University School of Medicine. The goal of the survey is to understand what adults think about CBD advertisements and will take about 15 minutes to complete. We expect that about 3,200 people will complete the survey. Upon completion of the survey, you will be provided with compensation agreed upon with your panel. Your participation is completely voluntary. Refusing to participate or leaving the study will not result in any penalty or loss of benefits to which you are entitled. You may choose not to take part or you may leave the study at any time.

The risk of harm or discomfort that may happen as result of taking part in this research study is not expected to be more than in daily life or from routine physical or psychological examinations or tests. All research studies involve some risks. A risk to this study that you should be aware of is the potential breach of confidentiality, however, we will do our best to protect your confidential information. Efforts, such as coding research records, keeping research records secure, and only allowing authorized people to have access to research records will be made to keep your information safe. No reference to any individual participant will appear in reports, presentations, or publications that may arise from the study. Identifiers might be removed from the identifiable private information and, after such removal, the information could be used for future research studies or distributed to another investigator for future research studies without additional informed consent from you or your legally authorized representative.

You are not expected to receive any direct benefit from taking part in this research study. We hope the information learned from this study will benefit other people in the future. This study is not intended to provide treatment for any disease or condition. The alternative to participating in the study is to not participate.

If you have any technical questions or complaints about this survey's functionality, or problems with incentives, please email AmeriSpeak at <a href="mailto:support@AmeriSpeak.org">support@AmeriSpeak.org</a> or call AmeriSpeak toll-free at 888-326-9424.

If you have any other questions, regarding this survey, or if you wish to withdraw from the study, please contact the study team at <a href="mailto:cbdresearch@wakehealth.edu">cbdresearch@wakehealth.edu</a>. If you have questions about your rights as a volunteer in this research, please contact the Wake Forest University School of Medicine Institutional Review Board at <a href="mailto:cbdresearch@wakehealth.edu">cbdresearch@wakehealth.edu</a>. If you have questions about your rights as a volunteer in this research, please contact the Wake Forest University School of Medicine Institutional Review Board at <a href="mailto:cbdresearch@wakehealth.edu">cbdresearch@wakehealth.edu</a>. If you have questions about your rights as a volunteer in this research, please contact the Wake Forest University School of Medicine Institutional Review Board at <a href="mailto:cbdresearch@wakehealth.edu">cbdresearch@wakehealth.edu</a>.

Checking the CONTINUE box below indicates that:

- You have read the above information
- You voluntarily agree to participate
- You are at least 18 years of age
- You authorize the use and disclosure of your health information as described in this consent and authorization form
- You understand that by taking part in this study, you are not releasing or agreeing to release the investigator, the sponsor, the institution or its agents from liability for negligence

| | _ | • |
|---------------------------------------------------|----|---|
| Check "CONTINUE" if you would like to participate | e: | |
| □ Continue | | |

□ EXIT